CLINICAL TRIAL: NCT01322646
Title: A Randomized Trial of Interventions for Teenage Drivers With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Gregory Fabiano, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD058588
Record Dates: First submitted 2010-08-11; First posted 2011-03-24 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Driving; Behavior modification
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Driver Training (Active Comparator): Driver Education Program Practice driving on a driving simulator Provision of the CarChipPro to the family
  Interventions: Device: CarChipPro; Behavioral: Driver's Education; Other: Driving Simulator Practice
- STEER Program (Experimental): Driver Education STEER Program
  Interventions: Device: CarChipPro; Behavioral: Driver's Education; Behavioral: STEER Program; Other: Driving Simulator Practice

INTERVENTIONS:
Device: CarChipPro — On board driving monitor
Behavioral: Driver's Education — 10 Session License to Learn Program.
Behavioral: STEER Program — 8-session behavioral parent training and teen social skills/communication training program
  Arms: STEER Program
Other: Driving Simulator Practice — Practice Driving on a driving simulator

SUMMARY:
There is clear, converging evidence from multiple prospective studies with well-diagnosed adolescents with ADHD and comparison, non-ADHD adolescents, that teen drivers with ADHD have more accidents and other adverse driving outcomes. Available research indicates parental monitoring and limit-setting for adolescent drivers is one of the most effective interventions for preventing negative driving outcomes. For children with ADHD, interventions to promote parenting capacity to effectively oversee and intervene in teen driving will likely need to be intensive and require multiple treatment components. The present proposal aims to compare the standard care for teen drivers (driver's education classes and driving practice) to the Supporting a Teen's Effective Entry to the Roadway (STEER) program, that includes a parent-teen intervention, adolescent skill building, parent training on effective adolescent management strategies, joint parent-teen negotiations sessions, practice on a driving simulator, parental monitoring of objective driving behaviors, and the targeting of safe teen driving via contingency management strategies (i.e., parent-teen contracts). To facilitate teen and parent engagement the intervention will be preceded by a motivational interview. The specific aims of the proposal are to investigate the efficacy of the STEER program relative to a standard care group in a randomized clinical trial (N=172) on measures of objective driving outcome and parenting capacity. It is hypothesized that the STEER program will result in improved outcomes relative to the standard care group at the end of intervention and 6 and 12 month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of ADHD, Combined Type
* At least 16 years old
* Has a driving Permit

Exclusion Criteria:

* No parent willing to be involved
* Seizure disorder, eating disorder, psychotic disorder, current diagnosis of substance/alcohol dependence
* Prior Driver's education class

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fabiano, PhD, Principal Investigator — SUNY at Buffalo
Locations (1):
- SUNY at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Result] Fabiano GA, Schatz NK, Morris KL, Willoughby MT, Vujnovic RK, Hulme KF, Riordan J, Howard M, Hennessy D, Lewis K, Hawk L, Wylie A, Pelham WE. Efficacy of a family-focused intervention for young drivers with attention-deficit hyperactivity disorder. J Consult Clin Psychol. 2016 Dec;84(12):1078-1093. doi: 10.1037/ccp0000137. Epub 2016 Sep 12. PMID 27618640

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Driver Training | STEER Program
Started | 86 | 86
Completed | 83 | 84
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Driver Training | STEER Program | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 86 | 172
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.88 (.65) | 16.98 (.7) | 16.92 (.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 61 | 63 | 124
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 86 | 172

OUTCOME MEASURES:

1. Primary Outcome: Number of Risky Driving Events Assessed by On-Board Driving Monitor
Description: Frequency count of risky driving events (e.g., abrupt braking, hard acceleration, abrupt swerving) recorded by engine performance monitor installed in the car. Events were counted and a greater frequency indicated more risky driving. The average number of risky driving events, collected over a four-week period at each assessment point were used as the dependent measure.
Time Frame: Follow up period after the intervention (1 year)
Measure: Least Squares Mean (Standard Error); unit: events
Arm/Group | Driver Training | STEER Program
Number analyzed (Participants) | 84 | 83
events | 3.20 (.58) | 3.95 (.73)

2. Primary Outcome: Positive Parenting Observational Data
Description: Parents and teens discussed two recent issues and these discussions were coded using The Interaction Behavior Code (IBC). The IBC is a behavioral coding system designed to assess global impressions of parent-adolescent problem-solving and communication behavior. Coders were undergraduates who were unaware of both study hypothesis and group assignment. Coders were instructed to rate 32 behavioral items related to positive and negative parenting in terms of their presence or absence of the behaviors (Items 1-22) or the how often specific parenting behaviors occurred for Items 23-32 ("no" = 0 points, "a little" = .5 point, and "alot" = 1 point). Coders scores were summed across the 32 items and scores fore each scale could range from 0-32. Thus for the positive parenting scale, higher scores, ranging from 0-32, indicated improvement.
Time Frame: Follow-up period after the intervention (12 weeks)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Driver Training | STEER Program
Number analyzed (Participants) | 84 | 83
score on a scale | .46 (.01) | .44 (.01)

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Arm/Group | Driver Training | STEER Program
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No